CLINICAL TRIAL: NCT03308812
Title: Impact of Technology-based Intervention for Improving Self-management Behaviors in Black Adults With Poor Cardiovascular Health: MECA Clinical Intervention Project
Brief Title: The Morehouse-Emory Cardiovascular Center for Health Equity Study: Clinical Intervention Project
Acronym: MECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00083584
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular health; Health coach; Cardiovascular risk factors; Ethnic disparities; Behavioral intervention; E-health lifestyle intervention; Health360x; eHealthyStrides
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health360x (Active Comparator): Participants will use the Health360x application for 6 months.
  Interventions: Behavioral: Health360x
- Health360x plus health coach (Experimental): Participants will use the Health360x application and received personalized health coaching for 6 months.
  Interventions: Behavioral: Health360x; Behavioral: Health Coach

INTERVENTIONS:
Behavioral: Health360x — Participants will view an orientation video which will include information on how to access the program from home and other internet access sites, how to use their activity monitor and sphygmomanometers, introduction to the curriculum, quizzes and discussion boards. Participants will be encouraged to upload their data at least once a week and to access the curriculum as often as desired. Technological and customer service support related to use of the application will be available 24 hours by phone.
  Other Names: eHealthystrides
Behavioral: Health Coach — Participants will be contacted by the health coach in the first week of the study to review their initial self-management behavioral goals and approaches. Follow up calls will occur each week for the first month, biweekly for the second and third months, and then once per month for the remainder of the study (months 4-6).
  Arms: Health360x plus health coach

SUMMARY:
This study will recruit from participants in the Morehouse-Emory Cardiovascular (MECA) study for a clinical intervention examining cardiac outcomes between participants who are randomized to received Health360x (a web-based and mobile-based application) or Health360x plus personalized health coaching. Participants will receive instruction on using the Health360x application and will use Health360x alone or Health360x with a health coach for 6 months. Measures of cardiovascular health will be assessed at baseline and after the 6 month long intervention.

DETAILED DESCRIPTION:
The internet can be an effective tool for driving behavior change but minority populations are less likely to engage or use this tool effectively. Health information technology (also called ehealth or e-health) can provide continuous and systematic connections to patients that will support their personal roles and responsibilities in their health care management. Ehealth technology allows for the tailoring of tools to the individual, timely information delivery, standardized messaging, layered content for more motivated participants, and the potential for greater efficiency/cost savings. Ehealth is able to provide effective and sustainable self-management tools for patients with chronic diseases. There is a significant trend towards information seeking on the internet among populations that have lower health literacy and are less trusting of the health system but, although minority and health disparities populations have increasing access to wireless and mobile technology, this has not translated to increased use of ehealth technologies.

The ehealth application used in this study aims to use the internet to engage vulnerable populations in improving their cardiovascular health. The intervention uses an enriched information environment, dynamic, personalized feedback on relevant health parameters, and social networks to impact health literacy, optimism and other resilience factors. This study will test two approaches to engagement with a robust ehealth application (Health360x) for high risk minority patients who reside in resilient and at risk neighborhoods within metro Atlanta. The Health360x application is a system that frames behavior as changeable and adaptable in a bidirectional manner, based on the behavioral constructs of Capability, Opportunity, and Motivation. Capability is the psychological and physical capacity to engage in the activity concerned, including the necessary knowledge and skills. Opportunity refers to factors that lie outside the individual, that facilitate or prompt the behavior. Motivation is largely governed by the brain processes that energize and direct behavior, including goal directed conscious decision-making, habitual processes, emotional response, as well as analytical decision-making.

This study is part of a larger project that is a partnership between investigators at Emory University and Morehouse School of Medicine who are actively involved in investigating ethnic disparities and incorporating the role of resilience factors in improving health status among black persons in metro Atlanta. The aim of this multi-disciplinary team is to establish a unique cohort in order to examine the associations between personal factors (psychosocial factors, socio-economic class, healthy behaviors and health beliefs) and environmental influences (neighborhood) on health behaviors and physiologic measures.

Four hundred subjects from "at risk" and "resilient" census tracks in metro Atlanta who completed the population surveys will be invited to participate in the Baseline Clinical Study, which is part of the Morehouse-Emory Cardiovascular (MECA) Center for Health Equity Study. The clinical trial described here will recruit 150 participants from the MECA study for a clinical intervention examining cardiac outcomes between participants who are randomized to received Health360x (a web-based and mobile-based application) or Health360x plus personalized health coaching.

Participants will receive instruction on using the Health360x application and will use Health360x alone or Health360x with a health coach for 6 months. Measures of cardiovascular health will be assessed at baseline and after the 6 month long intervention.

ELIGIBILITY:
Inclusion Criteria:

* Already participating in the Baseline Clinical Study
* Life Simple 7 (LS7) score of 8 or lower
* Internet access
* Self-reported ability to participate in physical activity
* English fluency

Exclusion Criteria:

* Coronary Artery Disease (CAD) documented by CAD diagnosis or prior acute myocardial infarction, percutaneous coronary intervention, coronary artery bypass surgery, or chronic angina
* Aortic stenosis
* History of chronic diseases that may alter brachial artery flow-mediated vasodilation measurements, such as peripheral vascular disease, HIV/AIDS, lupus, or cancer
* Inability to participate in increased physical activity
* History of alcohol or drug abuse or psychiatric diagnosis that would interfere with ability to participate
* Women who are pregnant and/or breastfeeding
* Cognitive deficits severe enough to preclude participation or any medical or surgical problem that precludes meaningful participation
* Unwillingness to use the internet

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Life Simple 7 (LS7) composite score | Baseline, Month 6
  The "Life Simple 7" (LS7) Cardiovascular Health Index is a public health metric by the American Heart Association (AHA) and is an index of modifiable health behaviors and cardiometabolic risk factors. The LS7 includes three health factors (blood pressure, fasting glucose, total cholesterol) and four health behaviors (body mass index (BMI), physical activity, healthy diet and smoking) and classifies each of them as "ideal" (score of 2), "intermediate" (score of 1) and "poor" (score of 0) levels. Total scores range from 0 to 14 and total scores between 0-4 are classified as inadequate, scores between 5-9 are considered average, and scores between 10-14 are classified as optimum cardiovascular health.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure | Baseline, Month 6
  Blood pressure readings will be made three times with the subject at rest in the sitting position using a cuff of the appropriate size and a standardized procedure. The average of the three systolic blood pressure measurements will be calculated. Blood pressure will be categorized according to Joint National Committee recommendations.
Change in Diastolic Blood Pressure | Baseline, Month 6
  Blood pressure readings will be made three times with the subject at rest in the sitting position using a cuff of the appropriate size and a standardized procedure. The average of the three diastolic blood pressure measurements will be calculated. Blood pressure will be categorized according to Joint National Committee recommendations.
Change in Delta Nutrition Intervention Research Initiative Food Frequency Questionnaire (Delta NIRI FFQ) | Baseline, Month 6
  Dietary intake of fruits and vegetables will be assessed using the Lower Mississippi Delta Nutrition Intervention Research Initiative food frequency questionnaire (Delta NIRI FFQ). The Delta NIRI FFQ is a 283-item, interviewer administered questionnaire that asks if respondents have had certain food items in the past 24 hours, including foods that are commonly consumed in the southern United States.
Change in Blood Glucose | Baseline, Month 3, Month 6
  Blood glucose will be measured as milligrams per deciliter at Baseline, 3 months after the start of the intervention and at the end of the intervention at month 6. Normal, fasting blood glucose levels are between 70 to 100 mg/dL.
Change in Distance Walked Daily | Baseline, Month 3, Month 6
  The total distance walked daily in miles will be measured by a pedometer or the exercise application for mobile devices.
Change in Short Form-12 Health Survey Questionnaire (SF-12) score | Baseline, Month 3, Month 6
  The Short Form-12 Health Survey Questionnaire (SF-12) is a measure of general physical and mental health. The SF-12 consists of 12 items with a Likert-type response format that measures quality of life with a Physical Component Summary (PCS) and Mental Component Summary (MCS). Subscales associated with the PCS include physical functioning, role limitations due to physical problems, bodily pain, and general health perceptions. Subscales associated with the MCS include vitality (energy and fatigue), social functioning, role limitations due to emotional problems, and mental health. The total score for each subscale ranges from 0 to 100 and low values represent a poor health state while high values represent a good health state.
Change in Stress Management | Baseline, then monthly through Month 6
  Participants will report on their stress management monthly via free text responses in an online format.
Change in Weight | Baseline, then monthly through Month 6
  Participants will report their weight in pounds once per month during the intervention period.
Change in Tobacco Use | Baseline, then monthly through Month 6
  Participants will report whether or not they have used tobacco once per month during the intervention period.

OTHER OUTCOMES:
Change in High-sensitivity C-reactive Protein (HsCRP) | Baseline, Month 6
  C-reactive protein (CRP) is a biomarker of cardiovascular health which increases in the blood when inflammation is present. The Hs-CRP test can measure low levels of CRP which indicate the risk of developing cardiovascular disease (CVD). A measurement of less than 1.0 milligrams of CRP per liter of blood (mg/L) is defined as low risk, 1.0 to 3.0 mg/L is average risk, and above 3.0 mg/L is high risk of developing CVD.
Change in Plasma Cysteine | Baseline, Month 6
  Plasma cysteine is a biomarker of oxidative stress, which is implicated in the pathophysiology of multiple conditions including cardiovascular disease (CVD). Higher levels of cysteine are associated with increased risk of CVD.
Change in Cystine | Baseline, Month 6
  Cystine is the oxidized form of cysteine. Higher plasma levels of cystine are associated with increased risk of CVD.
Change in CD34+ Cell Count | Baseline, Month 6
  Cells expressing CD34 antigen (a protein encoded by the CD34 gene) are called CD34+ cells and can be isolated from blood samples. CD34+ cell count is a biomarker of regenerative capacity and reduced counts of CD34+ is associated with increased cardiovascular risk.
Change in Pulse Wave Velocity (PWV) | Baseline, Month 6
  Carotid-femoral artery pulse wave velocity (PWV) will be determined using transcutaneous Doppler flow velocity recordings simultaneously over the common carotid artery and the femoral artery. Aortic pulse wave velocity (PWV) estimates of the speed of the pressure wave traveling along the aorta and is regarded as a direct measure of large artery stiffness. Normal ranges for PWV are age based (PWV increases with age) and standardized thresholds for CVD risk have not been established. This study will assess the change in PWV in participants between baseline and after the 6 month intervention.
Change in Reactive Hyperemia Index (RHI) | Baseline, Month 6
  Reactive Hyperemia Index (RHI) is a measure of microvascular endothelial function that is calculated as a ratio of preocclusion to postocclusion pulse signal amplitude. RHI will be estimated using digital pulse amplitude tonometry (EndoPAT). Greater RHI indicates better endothelial function.
Change in Glutathione | Baseline, Month 6
  Glutathione is a major antioxidant that helps eliminate peroxides and maintain cellular redox. Lower levels of glutathione are associated with cardiovascular disease.
Change in circulating progenitor cells (CPC) CD34+/CD133+ | Baseline, Month 6
  Progenitor cells (PCs), including CD34+/CD133+ cells, are part of the mechanisms underlying regeneration, and the pivotal role they play in vascular repair has only recently been appreciated. Endogenous PCs contribute to re-endothelialization of tissues after endothelial injury, attenuating progression to frank atherosclerosis. Endothelial dysfunction correlates with PC number and function and a low PC count appears to be an independent predictor of poor outcome in patients with CAD, stroke or acute lung injury. CD34+/CD133+ cell counts improved risk prediction metrics beyond standard risk factors.
Change in circulating progenitor cells (CPCs) CD34+/VEGF2R+ | Baseline, Month 6
  Progenitor cells (PCs), including CD34+/VEGF2R+ cells, are part of the mechanisms underlying regeneration, and the pivotal role they play in vascular repair has only recently been appreciated. Endogenous PCs contribute to re-endothelialization of tissues after endothelial injury, attenuating progression to frank atherosclerosis. Endothelial dysfunction correlates with PC number and function and a low PC count appears to be an independent predictor of poor outcome in patients with CAD, stroke or acute lung injury.
Change in Augmentation Index | Baseline, Month 6
  Augmentation index (AIx) is a composite measure of the magnitude of arterial wave reflections and systemic arterial stiffness and increases as the aortic pulse wave velocity (PWV) increases. Impaired arterial elastic properties, measured as the aortic AIx and/or PWV, are increasingly recognized as independent predictors of incident CVD events (myocardial infarction, stroke, revascularization), as well as all-cause mortality.
Change in Carotid Intima Media Thickness (CIMT) | Baseline, Month 6
  A CIMT scan is performed by using ultrasound determine the presence and severity of vascular disease. Presence of carotid plaque is associated with a 2-3-fold increased risk of future CVD events, and increased CIMT is associated with prevalent cardiovascular disease and an increased risk of myocardial infarction and stroke. Progression of CIMT has been used as a surrogate marker of change in CVD risk.

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Health System, Atlanta, Georgia
  - Morehouse School of Medicine, Clinical Research Center, Atlanta, Georgia
  - Emory University Clinical Research Network, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Islam SJ, Kim JH, Topel M, Liu C, Ko YA, Mujahid MS, Sims M, Mubasher M, Ejaz K, Morgan-Billingslea J, Jones K, Waller EK, Jones D, Uppal K, Dunbar SB, Pemu P, Vaccarino V, Searles CD, Baltrus P, Lewis TT, Quyyumi AA, Taylor H. Cardiovascular Risk and Resilience Among Black Adults: Rationale and Design of the MECA Study. J Am Heart Assoc. 2020 May 5;9(9):e015247. doi: 10.1161/JAHA.119.015247. Epub 2020 Apr 28. PMID 32340530